CLINICAL TRIAL: NCT03667820
Title: Phase II Trial of Osimertinib in Combination With Stereotactic Ablative Radiation (SABR) in EGFR Mutant Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Osimertinib and Stereotactic Ablative Radiation (SABR) in EGFR Mutant NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sawsan Rashdan, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122017-017
Record Dates: First submitted 2018-06-29; First posted 2018-09-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Osimertinib in combination with Stereotactic Ablative Radiation (SABR)
  Interventions: Drug: Osimertinib; Radiation: SABR

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 80mg tablet to be taken once daily.
  Other Names: AZD9291; TAGRISSO
Radiation: SABR — Stereotactic Ablative Radiation (SABR)

SUMMARY:
This study evaluates the combination of two well-tolerated therapies, osimertinib and Stereotactic Ablative Radiation (SABR).

DETAILED DESCRIPTION:
Patients with EGFR mutant non-small cell lung cancer will receive the current optimal therapy with osimertinib. After 8 weeks of targeted therapy, there will likely be some persisting lesions that would not have completely regressed. These persisting lesions would likely consist of cells that are less sensitive to targeted therapy. From the data summarized above [14], these persisting lesions are most to subsequently develop resistance and demonstrate progression.

To delay the onset of clinical progression, lesions that persist after 8 weeks of osimertinib therapy and are amenable to stereotactic ablative radiation will be radiated. Osimertinib will be held for 3 days before the first dose of radiation and resumed 3 days after the last dose.

After radiation, all patients will continue osimertinib therapy. If subsequently there is any evidence of progression, there will be an assessment of whether a repeat course of radiation is feasible. If it is feasible to repeat SABR to sites of progression, this will be performed and osimertinib resumed. If SABR is not possible, then a change in systemic therapy will be required.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent
* Age > 18 years
* Advanced EGFR exon 19 or 21 mutant NSCLC, not amenable to curative surgery or radiotherapy. EGFR mutations may be demonstrated by standard, clinically accepted methods, including direct gene sequencing, PCR, and NextGen sequencing.
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must have a life expectancy ≥ 12 weeks.
* Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Male patients should be willing to use barrier contraception.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* At least one lesion, not previously irradiated, that can be accurately assessed at baseline with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* Adequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count >1.5 x 109/L
  * Platelet count >100 x 109/L
  * Haemoglobin >9.0 g/dL (transfusion is permitted to achieve Hgb ≥9.0 g/dL)
  * Alanine aminotransferase <2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or <5 times ULN in the presence of liver metastases
  * Aspartate aminotransferase <2.5 times ULN if no demonstrable liver metastases or <5 times ULN in the presence of liver metastases
  * Total bilirubin <1.5 times ULN if no liver metastases or <3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
  * Serum Creatinine <1.5 times ULN concurrent with creatinine clearance >50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.

Exclusion Criteria

* Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site).
* Previous treatment with osimertinib or any EGFR TKI.
* Previous treatment with immunotherapy or any check point inhibitors.
* Treatment with an investigational drug within five half-lives of the compound
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 week prior) (Appendix A). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Patients with symptomatic CNS metastases who are neurologically unstable
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* History of hypersensitivity to osimertinib (or drugs with a similar chemical structure or class to osimertinib) or any excipients of these agents
* Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

In addition, the following is considered a criterion for exclusion from the exploratory genetic research:

* Previous allogeneic bone marrow transplant.
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Determine efficacy of Osimertinib plus SABR in patients with EGFR mutant lung cancer measured by Progression-Free Survival (PFS) | Every 8 weeks from the time of first dose of study medication until subject death from any cause, assessed up to 300 weeks.
  Progression-Free Survival (PFS) as determined by RECIST 1.1 or death (in the absence of progression).

SECONDARY OUTCOMES:
Determine the impact of Osimertinib plus SABR on survival | From time of first dose of study medication until subject death from any cause, up to 300 weeks.
  Overall survival defined as time from the date of initiation of Osimertinib until death of any cause.
Determine the impact of Osimertinib plus SABR on length of response | Every 8 weeks from time of first dose of study medication until disease progression or death from any cause, assessed up to 300 weeks.
  Duration of response (DoR) defined as the time from documentation of tumor response to disease progression.
Determine the impact of Osimertinib plus SABR on the length of time until next therapy needed | Every 8 Weeks from time of first dose of study medication until subsequent SABR, discontinuation, or disease progression, assessed up to 300 weeks.
  Time to subsequent SABR (2nd, 3rd, etc), initiation of new therapy, or death.
Determine the impact of Osimertinib plus SABR on tumor response | Every 8 weeks from time of first study medication dose until discontinuation or subject death from any cause, assessed up to 300 weeks.
  Objective response rate (ORR) defined as the proportion of patients with measurable disease who had a response after receiving at least one cycle of therapy.
Determine the impact of Osimertinib plus SABR on the duration of time while on Osimertinib | Every 8 weeks from time of first study medication dose until disease progression, discontinuation or subject death from any cause, up to 300 weeks.
  Impact defined as time from initiation of Osimertinib to evidence of disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason.
Number and type of adverse events related to Osimertinib plus SABR as assessed by CTCAE v4.0 | From time of first study medication dose through treatment period and including the follow-up period every 4 months following last dose of study medication, until subject death from any cause, up to 48 months.
  Defined as the risk to patients by using Osimertinib plus SABR and the degree to which overt adverse events of the Osimertinib plus SABR can be tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Sawsan Rashdan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sampath S, Rashdan S, Iyengar P, Mickel TA, Zhang S, Ahn C, Gao A, Dowell JE, Zhang Y, Westover KD, Cole SM, Amini A, Rock A, Massarelli E, Koczywas M, Gerber DE. Osimertinib plus consolidative radiotherapy for advanced EGFR mutant non-small cell lung cancer: a multicentre, single-arm, phase 2 trial. EClinicalMedicine. 2025 Aug 26;87:103435. doi: 10.1016/j.eclinm.2025.103435. eCollection 2025 Sep. PMID 41054436